CLINICAL TRIAL: NCT00842855
Title: Partial Response to PPI Treatment: The Cost to Society and the Burden to the Patient
Brief Title: Partial Response to PPI Treatment: The Cost to Society and the Burden to the Patient - a Study in France
Acronym: REMAIN
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: i3 Innovus (Industry)
Responsible Party: Debra Silberg, MD PhD, Medical Science Director, AstraZeneca R&D
Other Study IDs: D9120N00013
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2011-02-07 (Estimated); Status verified 2011-02

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD; PPI; partial responders
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: 274 GERD patients, partial responders to PPI treatment

SUMMARY:
The purpose of this study is to describe common treatment pathways, to collect health care utilization data and to assess symptom load as well as impact of symptoms on daily life in GERD patients who are partial-responders to PPI treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 month history of GERD symptoms
* Treated with unchanged optimized PPI treatment for any GERD indication during the last 4 weeks before enrollment
* Remaining GERD symptoms despite optimized PPI treatment
* Able to read and write in French, and able to comply with study requirements

Exclusion Criteria:

* Patients that have not experienced any GERD symptom improvement at all during PPI treatment
* Involvement in the planning or conduct of the study
* Involvement in any other observational study or in any clinical study at the time of this study or during the last 6 months
* Prior surgery of the upper GI tract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Gastroesophageal Reflux Disease (GERD) classified as partial responders to proton pump inhibitors (PPIs).
Sampling Method: Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Productivity loss; Frequency and severity of GERD symptoms; Health care resource use | Collected at enrollment visit and at 3, 6, 9 and 12 month follow-up. (Health care resource use is collected by the physician at enrollment visit and 6 and 12 month follow-up)
Utility values; Quality of Life | Collected at enrollment visit and at 6 and 12 month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Pr Stanislas Bruley des Varannes, MD PhD, Principal Investigator — Institut des Maladies de l'Appareil digestif; Marie Sundin, Study Director — AstraZeneca
Locations (44):
- France (44):
  - Research Site, Bandol
  - Research Site, Beaumont-sur-Oise
  - Research Site, Beausoleil
  - Research Site, Behren-lès-Forbach
  - Research Site, Berck
  - Research Site, Bièvres
  - Research Site, Bordeaux
  - Research Site, Bressuire
  - Research Site, Brest
  - Research Site, Cambrai
  - Research Site, Chalon-sur-Saône
  - Research Site, Colmar
  - Research Site, Cornebarrieu
  - Research Site, Creil
  - Research Site, Créteil
  - Research Site, Dieppe
  - Research Site, Freyming-Merlebach
  - Research Site, Gien
  - Research Site, Hagondange
  - Research Site, Ivoy-le-Pré
  - Research Site, La Garde
  - Research Site, La Rochelle
  - Research Site, La Seyne-sur-Mer
  - Research Site, Le Lavandou
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Mont-de-Marsan
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Rouen
  - Research Site, Saint-Cyr-sur-Mer
  - Research Site, Saint-Jeannet
  - Research Site, Saint-Mandé
  - Research Site, Saint-Mandrier-sur-Mer
  - Research Site, Sanary-sur-Mer
  - Research Site, Six-Fours-les-Plages
  - Research Site, Stiring-Wendel
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Toussieu
  - Research Site, Venerque
  - Research Site, Verdun
  - Research Site, Versailles
  - Research Site, Witry-lès-Reims